CLINICAL TRIAL: NCT01651312
Title: An Open-label Study to Evaluate the Pharmacokinetics of YM178 After Single Oral Administration of 14C-labeled YM178 in Healthy Male Volunteers
Brief Title: A Study to Assess the Systemic Pharmacokinetics, Metabolism and Excretion Routes of YM178 in Man, After Administration of Radio-labeled YM178
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-007
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Metabolic Processes
Keywords: Radioactivity; Excretion rate; Human subjects; Pharmacokinetics; YM178; Radio-labeled; Phase 1
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-labeled YM178 (Experimental): Single oral administration of 14C-labeled YM178
  Interventions: Drug: 14C-labeled YM178

INTERVENTIONS:
Drug: 14C-labeled YM178 — oral solution (1.85 MBq)
  Other Names: mirabegron; Myrebtriq

SUMMARY:
The study aims to assess the routes and the extent of metabolism and excretion of YM178 after a single dose of 14C-radiolabeled YM178 administered as a drinking solution in healthy male volunteers.

DETAILED DESCRIPTION:
Four subjects are studied in one group. Each subject stays in the clinic for 6 days, and receives a single oral dose of 14C-labeled YM178. Blood, plasma, urine, feces and expired air are collected for 96h after dosing.

If 14C-radioactivity quick counts show that radioactivity in urine or feces is above acceptable limits (ie. > 50 dpm/ml in urine; >75 dpm in 400 mg feces) on day 5, subjects are requested to stay in the clinic until the levels decrease. If, after 3 days, radioactivity is still > 50 dpm/ml in urine and/or >75 dpm in 400 mg feces, urine and/or feces is collected at home, until the amount of radioactivity decreases.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60 and 100 kg, and BMI ≤30 kg/m2

Exclusion Criteria:

* Known or suspected hypersensitivity to β-adrenergic receptor agonists or constituents of the formulations used
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug
* Any clinically significant history of upper gastrointestinal symptoms (such as nausea, vomiting, abdominal discomfort or upset, or heartburn) in the 4 weeks prior to admission to the Research Unit
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic
* Abnormal pulse rate measurement (<40 or >90 bpm) taken by manual counting at the pre-study visit after subject has been resting in supine position for 5 min
* Abnormal blood pressure measurements taken at the pre-study visit after subject has been resting in supine position for 5 min as follows:

  * Systolic blood pressure <95 or >160 mmHg;
  * Diastolic blood pressure <40 or >95 mmHg.
* Positive orthostatic test at screening i.e. any symptoms of dizziness, light-headedness etc. and/or a fall of ≥ 20 mmHg in systolic blood pressure after 2 min standing (preceded by 5 min. supine rest) and/or an increase in pulse rate of ≥ 20 bpm
* Regular use of any prescribed or OTC (over the counter) drugs except paracetamol up to 3 g/day, in the 4 weeks prior to admission to the Research Unit OR any use of such drugs in the 2 weeks prior to admission to the Research Unit
* History of drug abuse at any time, OR any use of drugs of abuse within 3 months prior to admission to the Research Unit
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Research Unit
* History of drinking more than 21 units of alcohol per week (1 unit = 270 cc of beer or 40 cc of spirits or 1 glass of wine) within 3 months prior to admission to the Research Unit
* Donation of blood or blood products within 3 months prior to admission to the Research Unit
* Positive serology test for HBsAg, HAV IgM, anti-HCV or anti-HIV 1+2.
* Participation in any clinical study within 3 months, or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study
* Subjects having received YM178 previously
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a clinical trial in the previous year

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2003-01; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
The assessment of pharmacokinetic profile of radioactivity after single-dose administration of 14C-YM178, measured by whole blood and plasma concentration | Baseline to Day 5 (optional (Day 6-8) [maximum of 19 assessments]
  Cmax, tmax, AUC0-last, AUC0-inf, t1/2 and the blood-to-plasma ratio (Ratio Cb/p)
The excretion rate and cumulative excretion of radioactivity in urine, feces and expired air after single-dose administration of 14C-YM178 | Baseline to Day 5 (optional (Day 6-8) [maximum of 10 assessments]
The assessment of pharmacokinetic profile of parent YM178 after single-dose administration of 14C-YM178, measured plasma and urine concentration | Baseline to Day 5 (optional (Day 6-8) [maximum of 19 assessments]
  plasma (Cmax, tmax, AUC0-last, AUC0-inf, t1/2 and Vz/F), urine (Ae0-24, Ae0-last, CLR and % dose excreted)

SECONDARY OUTCOMES:
Safety assessed through Adverse Events, vital signs, laboratory analyses and ECG (electrocardiogram) | Through to Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Pharma Bio-Research Group B.V., Zuidlaren, Netherlands

REFERENCES:
- [Background] Takusagawa S, van Lier JJ, Suzuki K, Nagata M, Meijer J, Krauwinkel W, Schaddelee M, Sekiguchi M, Miyashita A, Iwatsubo T, van Gelderen M, Usui T. Absorption, metabolism and excretion of [(14)C]mirabegron (YM178), a potent and selective beta(3)-adrenoceptor agonist, after oral administration to healthy male volunteers. Drug Metab Dispos. 2012 Apr;40(4):815-24. doi: 10.1124/dmd.111.043588. Epub 2012 Jan 23. PMID 22269146